CLINICAL TRIAL: NCT02928861
Title: 18F-FDG PET/CT-based Prognostic Model for Predicting Outcome in Patients With Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xuejuan Wang,MD, Department of Nuclear Medicine, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XW-DLBCL-002
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: Positron-Emission Tomography; Prognosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-FDG PET/CT-based prognostic model (Experimental): The new prognostic model is based on 18F-FDG PET/CT scans, and combined with clinical and pathological prognostic factors.
  Interventions: Device: 18F-FDG PET/CT

INTERVENTIONS:
Device: 18F-FDG PET/CT — 18F-FDG PET/CT will be conducted before, during and after chemotherapy. Patients were instructed to fast for at least 6 h before PET. The blood glucose level was measured to ensure that it was <200 mg/ dL. 18F-FDG was intravenously administered at a dose of 3.7 MBq/kg. Approximately 60 ± 10 min post- injection, a whole-body acquisition commenced in 6-8 bed positions (1 min/bed) using a hybrid system (PHILIPS Gemini TF) and covered from the base of the skull to the upper thigh, which was followed by CT in a non-contrast phase (modulated 100 mAs; 120 kV; slice thickness, 3 mm) for attenuation correction and anatomical localization purposes. The head acquisition was performed in one bed position (8-10 min/bed).

SUMMARY:
The purpose of this study is to evaluate whether 18F-FDG PET/CT-based prognostic model of diffuse large B-cell lymphoma can predict disease progression

DETAILED DESCRIPTION:
In this study investigators develop a prognostic model based on 18F-FDG PET/CT and test its ability for prognostic value in patients with DLBCL. PET/CT scans evaluation using the liver SUVmax as reference. Positive lesions in PET were indicated as SUVmax of residues higher than the threshold (1.6 fold of liver SUVmax) or new 18F-FDG avid lesions. 18F-FDG PET/CT-based prognostic model includes PET/CT image, dominant clinical and pathological prognostic factors to predicting disease progression during chemotherapy or survival in DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed DLBCL;
2. treated using an anthracycline-containing regimen with or without rituximab;
3. minimal follow-up at 6 months after the completion of first-line treatment;
4. complete medical history and clinicopathological data

Exclusion Criteria:

1. secondary malignant disease;
2. serious infection or inflammation (e.g., HIV);
3. primary central nervous system lymphoma;
4. hepatic or renal dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
2 year progression-free survival | up to 2 years after initial diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Xuejuan Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan T, Chen X, Zhang Y, Wei M, Zhu H, Yang Z, Wang X. A novel prognostic index for diffuse large B-cell lymphoma combined baseline metabolic tumour volume with clinical and pathological risk factors. Nucl Med Commun. 2023 Jul 1;44(7):622-630. doi: 10.1097/MNM.0000000000001701. Epub 2023 Apr 28. PMID 37114393
- [Derived] Yuan T, Zhang Y, Chen X, Wei M, Zhu H, Song Y, Yang Z, Zhu J, Wang X. Risk Assessment in Diffuse Large B-Cell Lymphoma by Combining Baseline Metabolic Tumor Volume and Peking Criteria When Evaluating Series 18F-Fluorodeoxyglucose Positron Emission Tomography Scans. Front Oncol. 2022 Apr 21;12:876581. doi: 10.3389/fonc.2022.876581. eCollection 2022. PMID 35530320